CLINICAL TRIAL: NCT04283084
Title: Development of Enhanced Virtual Reality Based Balance and Coordination Training System and Evaluation of Its Effectiveness
Brief Title: Development and Evaluation of Balance and Coordination Training System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09.2017.257
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Healthy; Coordination and Balance Disturbances; Lower Extremity Problem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Number of participants in this group is anticipated to be 25. Participants in this group will be receiving 10 minutes of exercise with the virtual reality based balance and coordination training system (MARBES). In the MARBES system two exercises (1. Balance exercise, 2. Coordination exercise) will be played for 5 minutes each.
  Interventions: Device: Virtual Reality Based Balance and Coordination Exercises

INTERVENTIONS:
Device: Virtual Reality Based Balance and Coordination Exercises — With the developed virtual reality based balance and coordination training system, balance and coordination exercises will be applied twice a week (12 sessions in total) for 6 weeks.

SUMMARY:
This project aims to develop an interactive floor that will perceive the pressure, give the user visual (light) and auditory (signal) feedback, use a monitor that will guide the user with visual reporting, develop a software that enables the integration of the floor with the monitor, adjusts the degree of difficulty of education, records training, and objectively grades balance development, investigate the clinical effectiveness of the balance and coordination education system, in which hardware and software coexist, verify the validity and reliability of the developed system by evaluating its validity and reliability with proven tests.

DETAILED DESCRIPTION:
In order to carry out daily life activities, independence of individuals should be insured. For this independence, it is necessary to have adequate balance and coordination. Without adequate balance and coordination, it is not possible to walk neither even to stand. Movement is the basic living unit of an organism. Balance and coordination are of great importance for smooth, fluid and convenient action. In the clinical settings individuals are given exercises in different ways to increase their balance and coordination to protect them from injuries and to gain their independence. Nowadays, in order to adapt to the future, technological devices that can analyze and improve balance and coordination are being developed. The adequacy of the devices or systems developed for this purpose is also discussed. Most of the systems available on market only provide balance training by moving the floor, while others aim to contribute to balance by stimulating joint proprioception with a vibrating ground. This project aims to develop equipments that will provide balance and coordination trainings to guide the user through visual, auditory and mechanical feedback, develop a software which will record, analyze and evaluate the trainings given while ensuring that this equipment works systematically, carry out clinical studies to investigate the effectiveness of this developed system in healthy people.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate
* Being healthy
* Being between 18-45 years of age

Exclusion Criteria:

* Presence of any neurological or orthopedic problems that may affect balance and coordination,
* Being pregnant,
* Any drug use that may affect balance and coordination,
* Any deformation in vertebrae or lower limbs,
* History of any surgery in the lower limbs in the preceding 1 year,
* Any nervous lesion, existing neurological diseases, sensory defects,
* Any hearing or visual problems

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-05-20 (Estimated); Study Completion 2021-06-20 (Estimated)

PRIMARY OUTCOMES:
Change in Y Balance Test from baseline to week 6 | 6 weeks
  The Y Balance Test (YBT) is a simple, yet reliable, test used to measure dynamic balance (1). It was developed to standardize the modified Star Excursion Balance Test (mSEBT), improve its practicality, and make it commercially available. The YBT requires the athlete to balance on one leg whilst simultaneously reaching as far as possible with the other leg in three separate directions: anterior, posterolateral, and posteromedial. Therefore, this test measures the athlete's strength, stability and balance in various directions. The YBT composite score is calculated by summing the 3 reach directions and normalizing the results to the lower limb length.
Change in Single-Leg-Stance Test from baseline to week 6 | 6 weeks
  The Single-Leg-Stance Test (SLST) is a static balance test that has been used widely in older adults and has normative data accepted by the scientific literature. To perform the test, the patient is instructed to stand on one leg without support of the upper extremities or bracing of the unweighted leg against the stance leg. The patient begins the test with the eyes open, practicing once or twice on each side. The patient is then instructed to close his eyes and maintain balance for up to 45 seconds. The number of seconds that the patient/client is able to maintain this position is recorded. Termination or a fail test is recorded if 1) the foot touches the support leg; 2) hopping occurs; 3) the foot touches the floor, or 4) the arms touch something for support.
Change in Lower Extremity Motor Coordination Test (LEMOCOT) from baseline to week 6 | 6 weeks
  The LEMOCOT consists of moving the lower extremity as fast as possible from 1 target to another for 20 seconds. The number of on-target touches constitutes the score.
Change in Pedalo Sensamove Balance Test from baseline to week 6 | 6 weeks
  Pedalo®-Sensomove balance device consists of a mini board which is a circular board with hemispheric shaped sensors placed below it and works as three-dimensional accelerometer and gyroscope with a sample frequency of 100 Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Dilara Merve Sari, MSc, Principal Investigator — Marmara University Institute of Health Sciences; Tugba Kuru Colak, PhD, Study Director — Marmara University Faculty of Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldie PA, Bach TM, Evans OM. Force platform measures for evaluating postural control: reliability and validity. Arch Phys Med Rehabil. 1989 Jul;70(7):510-7. PMID 2742465
- [Background] Desrosiers J, Rochette A, Corriveau H. Validation of a new lower-extremity motor coordination test. Arch Phys Med Rehabil. 2005 May;86(5):993-8. doi: 10.1016/j.apmr.2004.11.007. PMID 15895347
- [Background] Woollacott M, Shumway-Cook A. Attention and the control of posture and gait: a review of an emerging area of research. Gait Posture. 2002 Aug;16(1):1-14. doi: 10.1016/s0966-6362(01)00156-4. PMID 12127181